CLINICAL TRIAL: NCT07296406
Title: Exploring the Efficacy of Application Managing Somatic Symptoms Disorder & Medically Unexplained Symptoms (MUS) : A Pilot Study
Brief Title: App-Based Self-Management for Somatic Symptom Disorder and MUS: A Pilot Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jooyoung Oh, Clinical Associate Professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2024-0119
Record Dates: First submitted 2025-09-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Somatic Symptom Disorder

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, parallel assignment trial with two arms (intervention vs. waitlist). Participants in the intervention group will use the mobile application for 8 weeks (V1-V2) followed by a 8-week follow-up period without app use (V2-V3). Participants in the waitlist control group will receive usual care for the first 8 weeks (V1-V2), and then begin using the mobile application for 8 weeks (V2-V3).
Masking Description: Open-label trial; no masking of participants, care providers, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Intervention Group (Experimental): Participants in this group will use the mobile self-management application for somatic symptom disorder and medically unexplained symptoms for 8 weeks, in addition to receiving their usual care.
  Interventions: Behavioral: Arm I (App Intervention); Behavioral: Arm II (Waitlist Control)
- Waitlist Control Group (No Intervention): Participants in this group will continue treatment as usual for 8 weeks without access to the mobile application. After the primary 8-week period, they will be offered access to the application.

INTERVENTIONS:
Behavioral: Arm I (App Intervention) — Participants assigned to the intervention group will use a mobile self-management application designed for individuals with somatic symptom disorder and medically unexplained symptoms. The app delivers psychoeducation, CBT- and mindfulness-based therapeutic content, stress management tools, and behavioral monitoring over a 8-week period, in addition to participants' usual care.
  Arms: App Intervention Group
Behavioral: Arm II (Waitlist Control) — Participants in the control group will continue treatment as usual for 8 weeks without access to the mobile application. After completion of the 8-week primary endpoint, they will be offered access to the mobile application.
  Arms: App Intervention Group

SUMMARY:
Objectives The primary objective of this study is to evaluate the effectiveness of an eight-week self-management mobile application for adults experiencing somatic symptom disorder (SSD) or medically unexplained symptoms (MUS). Improvement will be assessed using the PHQ-15. The secondary objective is to examine changes in clinical symptoms and physiological indicators following app use, as well as to assess the acceptability and usability of the intervention.

Scientific Rationale Somatic symptoms without clear medical explanation account for 15-30% of primary care visits (Peveler et al., 1997; Fink et al., 1999; Ko et al., 2011). Diagnostic terminology has evolved from somatoform disorders in DSM-IV and MUS to SSD in DSM-5, which emphasizes distressing symptoms accompanied by maladaptive thoughts, emotions, or behaviors (Scott et al., 2022). SSD is frequently associated with alexithymia, emotional suppression, and difficulty regulating anger, consistent with theories of somatization as the bodily expression of unprocessed affect (Anuk & Bahadir, 2017; Liu et al., 2011). These difficulties contribute to interpersonal impairment and excessive health care use, often resulting in frustration for clinicians (Orzechowska et al., 2020).

Psychological treatments, including CBT, MBSR, MBCT, and ACT, have demonstrated efficacy in reducing symptom burden across conditions such as IBS, fibromyalgia, tinnitus, and chronic fatigue (Hauge et al., 2015; Kikuchi et al., 2020; Roland et al., 2015). These therapies share mechanisms such as enhancing mind-body awareness, reducing physiological hyperarousal, and promoting adaptive coping and acceptance (Aktas et al., 2019; Jing et al., 2019). However, barriers to dissemination remain, as patients with SSD often reject psychological explanations, engage in medical shopping, and maintain strong somatic attributions (Brown, 2007; Harris et al., 2009).

Digital interventions offer a scalable solution by providing psychoeducation on mind-body connections, CBT- and mindfulness-based strategies, stress management tools, and behavioral monitoring in an accessible, daily-life format. Evidence suggests that internet- and app-based CBT programs can improve somatic distress and related outcomes, while also reducing treatment costs and improving adherence (Van et al., 2022).

Physiological measures such as heart rate variability (HRV) provide an objective biomarker of stress regulation. Lower HRV reflects reduced resilience and greater emotional dysregulation, while higher HRV indicates excessive arousal or impaired recovery. Despite theoretical links between autonomic regulation and somatization, few studies have examined HRV responses in SSD populations alongside psychological interventions. This study addresses that gap.

Study Design A randomized controlled trial will recruit 110 adults aged ≥19 years who report significant somatic distress. After screening and informed consent, participants will be randomly assigned (1:1) to intervention (n=55) or control (n=55) using an R-generated allocation table managed independently of investigators.

Baseline assessments include standardized questionnaires and HRV measurement. The intervention group will use the mobile application for eight weeks, while the control group will continue treatment as usual. After eight weeks, both groups will complete follow-up questionnaires and HRV measurement. Subsequently, the intervention group will discontinue app use, and the control group will be offered app access. An additional follow-up survey will be conducted online for both groups at 16 weeks.

Expected Impact This study will provide empirical evidence on the efficacy, usability, and acceptability of a digital intervention for SSD and MUS. By integrating self-management strategies with physiological monitoring, it aims to advance scalable, evidence-based approaches for a population that has historically been difficult to treat within traditional medical models.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* PHQ-15 score of 4 or higher
* Presence of medically unexplained physical symptoms (MUS)
* No significant impairment in reading or writing ability
* Familiarity with smartphone and internet use

Exclusion Criteria:

* Current diagnosis of substance use disorder (alcohol or drugs)
* Current diagnosis of schizophrenia or bipolar disorder, or presence of psychiatric symptoms deemed by the clinician to interfere with participation
* Currently receiving psychotherapy specifically for somatic symptoms
* Diagnosis of developmental disorders such as autism or intellectual disability, or evidence of significant cognitive impairment
* Any other medical condition deemed by the clinician to make participation inappropriate
* Inability to continue participation due to smartphone malfunction or lack of sufficient smartphone skills

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Somatic Symptom Severity (Patient Health Questionnaire-15; PHQ-15) | Baseline, 8 weeks after intervention start (V2), 16 weeks after intervention start (V3)
  The primary outcome is the change in somatic symptom severity measured by the Patient Health Questionnaire-15 (PHQ-15). The PHQ-15 is a 15-item self-report scale developed to assess the severity of somatic symptoms in primary care (Kroenke et al., 1998) and validated in psychiatric outpatient populations (Han et al., 2009). Scores range from 0 to 30, with higher scores indicating greater somatic symptom burden.

SECONDARY OUTCOMES:
Somatic Symptom Disorder B-Criteria Scale (SSD-12) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Somatic symptom-related cognitive, affective, and behavioral distress will be assessed using the Somatic Symptom Disorder B-Criteria Scale (SSD-12). The SSD-12 is a 12-item self-report measure that evaluates the psychological B-criteria of somatic symptom disorder, including excessive health-related thoughts, negative emotions, and maladaptive behaviors in response to somatic symptoms. Each item is rated on a 0-4 scale, with higher scores indicating greater somatic symptom-related psychological distress.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Depressive symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report scale that assesses the frequency of core depressive symptoms over the past week, with items rated from 0 ("not at all") to 3 ("nearly every day"). Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item self-report questionnaire that measures the severity of generalized anxiety symptoms over the past week, with each item rated from 0 ("not at all") to 3 ("nearly every day"). Total scores range from 0 to 21, with higher scores indicating greater anxiety severity.
Liebowitz Social Anxiety Scale, Self-Rated (LSAS-SR) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Social anxiety symptoms will be measured using the self-rated version of the Liebowitz Social Anxiety Scale (LSAS-SR). The LSAS-SR consists of 20 items assessing fear and avoidance across a range of social and performance situations, with each item rated on 0-4 scales for fear and avoidance. Higher scores reflect more severe social anxiety and greater avoidance of social situations.
Korean Version of the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Trait mindfulness will be assessed using the Korean version of the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF). The FFMQ-SF is a 15-item self-report scale that evaluates five facets of mindfulness: non-reactivity, observing, acting with awareness, describing, and nonjudging. Items are rated on a 1-7 scale, with higher scores indicating higher levels of dispositional mindfulness across these facets.
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Psychological acceptance will be measured using the Korean version of the Acceptance and Action Questionnaire-II (AAQ-II). The AAQ-II is a self-report measure that assesses acceptance of internal experiences and willingness to act in line with values in the presence of difficult thoughts and feelings. Items are rated on a Likert-type scale, and in the Korean scoring used in this study, higher scores indicate a higher level of acceptance and openness toward internal experiences.
Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Cognitive emotion regulation strategies will be assessed using the Cognitive Emotion Regulation Questionnaire (CERQ). The CERQ is a 35-item self-report measure that evaluates nine cognitive strategies used in response to negative life events, including acceptance, putting into perspective, positive refocusing, refocus on planning, positive reappraisal, self-blame, catastrophizing, other-blame, and rumination. Items are rated on a 1-5 scale, with higher subscale scores indicating more frequent use of the corresponding cognitive emotion regulation strategy.
Intolerance of Uncertainty Scale - Short Form (IUS-12) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Intolerance of uncertainty will be measured using the 12-item Intolerance of Uncertainty Scale - Short Form (IUS-12). The IUS-12 assesses negative beliefs, distress, and difficulty functioning in situations involving ambiguity or uncertainty, with items rated on a 1-4 scale. Higher scores indicate greater intolerance of uncertain or ambiguous situations.
Forms of Self-Criticism/Attacking and Self-Reassuring Scale (FSCRS) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Self-criticism and self-reassurance will be assessed using the Korean version of the Forms of Self-Criticism/Attacking and Self-Reassuring Scale (FSCRS). The FSCRS is an 18-item self-report measure that assesses two main dimensions: self-critical attitudes and self-reassuring responses toward oneself when facing setbacks or failures. Items are rated on a 0-4 scale, with higher scores on self-criticism indicating more frequent self-attacking, and higher scores on self-reassurance indicating a greater ability to respond to oneself with kindness and support.
Illness Attitudes Scale (IAS) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Health-related attitudes and concerns will be measured using the Illness Attitudes Scale (IAS). The IAS is a 27-item self-report scale that assesses hypochondriacal concerns, health anxiety, disease conviction, and related illness attitudes. Items are rated on a 0-4 scale, with higher scores reflecting more negative or maladaptive attitudes and fears related to illness.
Korean Multidimensional Assessment of Interoceptive Awareness (K-MAIA) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Interoceptive awareness will be assessed using the Korean Multidimensional Assessment of Interoceptive Awareness (K-MAIA). The K-MAIA is a 32-item self-report scale that measures multiple dimensions of how individuals perceive and relate to internal bodily sensations, including noticing, attention regulation, emotional awareness, self-regulation, and body listening. Items are rated on a 0-5 scale, with higher scores indicating more adaptive and accurate interoceptive awareness.
Korean Shapiro Control Inventory (K-SCI; Control and Desire for Control Subscales) | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Perceived control and desire for control will be measured using the Korean version of the Shapiro Control Inventory (K-SCI), focusing on the positive control, negative control, and desire for control subscales. These subscales together comprise 24 items rated on a 1-7 scale and assess individuals' beliefs about their ability to exert control, their experiences of lacking control, and their motivation to maintain or increase control. Higher scores on each subscale indicate stronger positive sense of control, greater negative control experiences, or greater desire for control, respectively.
App Usability and Acceptability | Baseline, 8 weeks after intervention start, and 16 weeks after intervention start
  Perceived usability and acceptability of the mobile application will be assessed using a 24-item self-report questionnaire adapted from prior work on smartphone-based interventions for serious mental illness. Items are rated on a three-point scale (disagree, neutral, agree) and evaluate ease of use, perceived usefulness, satisfaction, and willingness to continue using or recommend the app. Higher scores indicate greater perceived usability, acceptability, and perceived value of the digital intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No